CLINICAL TRIAL: NCT03568279
Title: Influence of Two-handed Jaw Thrust on Postoperative Sore Throat
Brief Title: Jaw-thrust on Postoperative Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JTPOST
Record Dates: First submitted 2018-06-04; First posted 2018-06-26 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The attending anesthesiologist provided intubation without two-handed jaw thrust.
  Interventions: Procedure: Control
- Two-hand (Experimental): The attending anesthesiologist provided intubation with two-handed jaw thrust.
  Interventions: Procedure: Two-handed jaw thrust

INTERVENTIONS:
Procedure: Two-handed jaw thrust — The assistant applied two-handed jaw thrust for intubation.
  Arms: Two-hand
Procedure: Control — The intubation was done without two-handed jaw thrust.
  Arms: Control

SUMMARY:
This investigation is planned to compare the incidence and severity of postoperative sore throat according to the use of two-handed jaw thrust maneuver in patients undergoing endotracheal intubation for general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients scheduled for general anesthesia with endotracheal intubation

Exclusion Criteria:

* Difficult airway
* Mallampatti scores greater than 2
* Recent sore throat
* Cervical spine disease
* Recent upper respiratory infection
* Recent analgesics
* History of head and neck surgery
* Friable teeth
* Multiple intubation attempts

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative sore throat for postoperative 24 hour | At postoperative 24 hour

SECONDARY OUTCOMES:
Number of participants with postoperative sore throat | At postoperative 2, 4, and 24 hour
Postoperative sore throat scores | At postoperative 2, 4, and 24 hour
  Visual analogue scales will be used (10: most imaginable pain, 0: no pain).
Number of participants with postoperative hoarseness | At postoperative 2, 4, and 24 hour
Number of participants with postoperative shivering | At postoperative 2, 4, and 24 hour
Wound pain scores | At postoperative 2, 4, and 24 hour
  Visual analogue scales will be used (10: most imaginable pain, 0: no pain).
Number of participants with jaw discomfort | At postoperative 2, 4, and 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Hyun-Chang Kim, Daegu, Non-US/Canada, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huh H, Go DY, Cho JE, Park J, Lee J, Kim HC. Influence of two-handed jaw thrust during tracheal intubation on postoperative sore throat: a prospective randomised study. J Int Med Res. 2021 Feb;49(2):300060520961237. doi: 10.1177/0300060520961237. PMID 33535830